CLINICAL TRIAL: NCT06257537
Title: Sustained Acoustic Medicine for Symptomatic Treatment of Knee Pain Related to Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KP-01-2024
Record Dates: First submitted 2024-02-02; First posted 2024-02-14 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Osteo Arthritis Knee; Arthritis
Keywords: Low-Intensity Ultrasound; Drug Delivery; Sonophoresis; Transdermal Drug Delivery; Non-Steroidal Anti-Inflammatory Drugs; Sustained Acoustic Medication; Low-Intensity Continuous Ultrasound
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- SAM Ultrasound Device and Diclofenac Patch (Experimental): Patients receive treatment from the wired SAM Ultrasonic Diathermy Device for 4 hours at least 5 days a week for 24 weeks combined with 2.5% diclofenac patch. The SAM Device emits continuous ultrasound at 3 megahertz(MHz) frequency and 0.132 watts/cm^2 intensity.
  Interventions: Device: Sustained Acoustic Device with 2.5% Diclofenac Patch
- SAM Ultrasound Device and SAM Patch (Active Comparator): Patients receive treatment from the wired SAM Ultrasonic Diathermy Device for 4 hours at least 5 days a week for 24 weeks combined with SAM patch (0% diclofenac).
  Interventions: Device: Sustained Acoustic Device with 0% Diclofenac Patch
- Diclofenac Patch (Active Comparator): Patients wear 2.5% diclofenac patch for 4 hours at least 5 days a week for 24 weeks combined.
  Interventions: Drug: 2.5% Diclofenac Patches
- SAM Patch (Placebo Comparator): Patients wear 0% diclofenac patch for 4 hours at least 5 days a week for 24 weeks combined.
  Interventions: Other: SAM Patch

INTERVENTIONS:
Device: Sustained Acoustic Device with 2.5% Diclofenac Patch — Patients apply the SAM Ultrasonic Diathermy Device daily for 1-4 hours of continuous therapeutic ultrasound at 3 megahertz(MHz) frequency and 0.132 Watts/cm^2 with 2.5% Diclofenac patches.
  Other Names: ZetrOZ Ultrasound Device; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS Device Wearable; Long Duration Low-Intensity Device
  Arms: SAM Ultrasound Device and Diclofenac Patch
Device: Sustained Acoustic Device with 0% Diclofenac Patch — Patients apply the SAM Ultrasonic Diathermy Device daily for 1-4 hours with 0% diclofenac patches.
  Other Names: ZetrOZ Ultrasound Device; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS Device Wearable; Long Duration Low-Intensity Device
  Arms: SAM Ultrasound Device and SAM Patch
Drug: 2.5% Diclofenac Patches — Topical pain relief-gel worn for 4 hours at least 5 days a week via SAM patch.
  Arms: Diclofenac Patch
Other: SAM Patch — Ultrasound gel without additional pain relief medication worn for 4 hours at least 5 days a week via SAM patch.
  Arms: SAM Patch

SUMMARY:
The purpose of this study is to assess the ability of long-duration low intensity therapeutic ultrasound (LITUS) to alleviate knee Osteoarthritis pain over a 24-week period.

The primary objective of this study is to evaluate the analgesic effect of LITUS in subjects suffering from knee Osteoarthritis pain.

Secondary objectives are to assess the ability of LITUS to improve joint function.

DETAILED DESCRIPTION:
This is a 24-week study to clinically evaluate the effectiveness of the wireless Sustained Acoustic Medicine (SAM) device combined with diclofenac on symptoms of patients suffering from knee osteoarthritis. The class-II device, sam®, has been FDA-cleared for home use. On the first day of the study, baseline data will be collected as patients report pain score before treatment. During the following 24 weeks, patients will self-apply their assigned treatment for the 4 hours daily. Each day of the study, pain scores will be recorded immediately before application of SAM device as well as at the completion of treatment. Assessments on quality of life & function, depression & anxiety, and sleep will be performed prior to the patient beginning the protocol, at 8 weeks, 16 weeks and at the conclusion of the protocol.

Over 300 subjects will be recruited from neighboring communities to the study sites. The study is designed to reach a target patient population which includes rural citizens and socioeconomic disadvantaged individuals.

ELIGIBILITY:
Inclusion Criteria:

* Have physician-diagnosed mild to moderate knee OA (OARSI atlas grades 1-2)
* Fulfill the American College of Rheumatology clinical and radiological diagnostic criteria for knee OA
* Are between 50-85 years of age
* Report a frequent pain score between 4-7 (range: 0-10) during the week preceding enrollment
* Report that knee pain negatively affects quality of life
* Are willing not to use any cream, gel, or topical solution during the administration of treatment other than the approved ultrasound gel provided to the subject at the initiation of the study
* Are deemed appropriate by their physician or by the study site physician to participate.
* Be willing and able to self-administer treatment daily within their place of residence or during normal daily activity, excluding bathing, showering, or other water activities which may result in submersion of the study device.
* Not use or initiate use of opioid and/or non-opioid analgesic medications.
* Be willing to discontinue any other interventional treatment modalities on the knee during the study period (e.g., transcutaneous electrical nerve stimulation, electronic muscle stimulation, traditional ultrasound).

Exclusion Criteria:

* Cannot successfully demonstrate the ability to put on and take off the device.
* Displays any condition which, in the judgment of the investigator, would make participation in the study unacceptable including, but not limited to, the subject's ability to understand and follow instructions.
* Participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening.
* Is pregnant.
* Is a prisoner.
* Is non-ambulatory (unable to walk).
* Has a pacemaker.
* Has a malignancy in the treatment area.
* Has an active infection, open sores, or wounds in the treatment area.
* Has impaired sensation in the treatment area, such as caused by chemotherapy or anesthesia.
* Has a known neuropathy (disease of the brain or spinal nerves).
* Has a hereditary disposition (tendency) for excessive bleeding (hemorrhage).
* Have knee replacement, other surgical intervention, or hyaluronidase injection in the affected knee in the past 6 months.
* Are currently taking steroids.
* Have any contraindication to radiograph.
* Have a secondary cause of arthritis (metabolic or inflammatory).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Units on a Scale (0-10) 0 Being Least, 10 Being Worst Pain From Baseline | Through study completion, average of 24 weeks.
  Change in the self-described pain units on a scale by patient at baseline and post-treatment.
Change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Through study completion, average of 24 weeks.
  WOMAC questionnaire will be utilized (Western Ontario and McMaster Universities Arthritis Index) at baseline and post-treatment to calculate the change in scores. WOMAC was divided into 3 categories: pain, stiffness, function and total score. The pain category consists of five scores from 0 - 4, 0 being no pain 4 is worst pain possible, for a range of 0 - 20 points. The stiffness category consists of two scores from 0 - 4, 0 being no stiffness 10 is worst stiffness possible for a range of 0 - 8 points. The function score consists of 17 scores from 0 - 4, 0 being normal function and 10 is severely limited function, for a range of 0 - 68 points. Total score is the sum of pain, stiffness, and function scores (range of 0 - 96).

SECONDARY OUTCOMES:
Change in Global Rating of Change (GROC) on a Scale (-7 to +7) | Through study completion, average of 24 weeks.
  Subject-reported change in overall pain on a scale, -7 = worst, +7 = best.
Change in the Pain & Sleep Questionnaire (PSQ-3) | Through study completion, average of 24 weeks.
  Subject-reported rating of impact of pain on sleep on a scale from 0 no impact, to 100 greatest impact.
Change in Depression Anxiety Stress Scale (DASS21) | Through study completion, average of 24 weeks.
  Subject-reported measures of depression, anxiety, and stress on a scale of 0-3, 0 being not applicable, 1 meaning applicable to some degree, 2 meaning applicable often, and 3 meaning applicable most of the time. Questions are divided into three categories: depression, anxiety, and stress.

CONTACTS AND LOCATIONS:
Overall Officials: George K Lewis, Ph.D., Principal Investigator — ZetrOZ Systems
Locations (3):
- United States (3):
  - Orthopaedic Foundation, Stamford, Connecticut
  - ZetrOZ Systems, Trumbull, Connecticut
  - Cayuga Medical Center - Medical Pain Consultants, Dryden, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Class II Medical Device — https://www.samrecover.com